CLINICAL TRIAL: NCT03286972
Title: PET/MRI to Enhance Precision Guidance in Head and Neck Radiation Treatment Planning
Status: Terminated | Type: Observational
Why Stopped: Slow accrual
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: UW16064; 2017-0162 (Other: Institutional Review Board); A533300 (Other: UW Madison); SMPH\HUMAN ONCOLOGY\HUMAN ONCO (Other: UW Madison); NCI-2019-05974 (Registry Identifier: NCI Trial ID)
Record Dates: First submitted 2017-09-14; First posted 2017-09-19 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-06

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PET/MRI: All participants will undergo a diagnostic PET/CT and a Radiation Treatment Planning CT per SOC procedures. In addition, all participants will undergo an additional imaging set consisting of a PET/MRI. It is anticipated that most patients will undergo the PET/MRI on the same day as their PET/CT negating the need for a second injection of the FDG radioisotope used for SOC PET imaging. All participants will receive gadolinium contrast per SOC dosing guidelines for the MRI portion of the PET/MRI. Both SOC MMRI pulse sequences and investigational sequences will be utilized in this study.
  If a second dose of the radioisotope is need to complete the PET/MRI (unable to perform both PET scans on the same day) only a 50% dose of FDG will be administered due to the increased sensitivity the PET/MRI scanner.
  Interventions: Device: PET/MRI

INTERVENTIONS:
Device: PET/MRI — Participants will be placed in standard non-ferrous head and neck immobilization devices during PET/MRI (to simulate their anticipated positioning during subsequent CT simulation and treatment). A head/neck PET/MRI (standard bore size, 60 cm) will be performed

SUMMARY:
The purpose of this study is to evaluate this new technology available at the University of Wisconsin Carbone Cancer Center in the setting of head and neck cancer radiation treatment planning. This study will also provide preliminary data critical to the development of multi-parametric, multi-modality quantitative imaging biomarkers and data analysis models for prediction of outcome in both tumors and normal tissue, which are essential for patient-specific adaptive therapy.

All participants will undergo a diagnostic PET/CT and a Radiation Treatment Planning CT per SOC procedures. In addition, all participants will undergo an additional imaging set consisting of a PET/MRI. It is anticipated that most patients will undergo the PET/MRI on the same day as their PET/CT negating the need for a second injection of the FDG radioisotope used for SOC PET imaging. All patients will receive gadolinium contrast per SOC dosing guidelines for the MRI portion of the PET/MRI. Both SOC MMRI pulse sequences and investigational sequences will be utilized in this study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with tumors of the head and neck region (nasal cavity, oral cavity, pharynx, larynx, sinuses, salivary glands, and head and neck skin) who are candidates for radiation treatment.

Exclusion Criteria:

* Contraindications for MRI: All patients will be screened with standard UWHC MRI screening procedures:
* Any person with the following will be excluded: cardiac pacemaker, metal fragments in or around the eye, venous umbrella, permanent eyeliner or permanent artificial eyebrows.

Patents with the following potentially non-MRI compatible devices will undergo screening using the standard UWHC MRI screening protocol by trained UWHC personnel: cardiac pacemaker, heart valve replacement, intracranial aneurysm clips, middle ear, eye, joint, or penile implants, joint replacements, implantable hearing aids, neurostimulator devices, insulin pumps, shunts/stents, metal mesh/coil implants; metal plate/pin/screws/wires, or any other metallic implants. Also patients with anatomical constraints limiting the feasibility of MRI will be excluded.

- Issue of pregnancy: We will exclude all known pregnant females from the study to avoid the potential risk of fetal injury upon exposure to the PET scan. Determination of pregnancy will be based upon the standard screening procedures in place for radiation therapy.

* Persons who are not fluent in English
* Anyone who can not provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The planned enrollment of 40 participants includes 4-12 patients in each of the 5 anatomic subgroups. This will allow flexibility in enrollment to reflect the frequency pattern of case presentation and any early findings that may suggest one or more sub-sites are particularly well suited to disclose valuable tumor data using PET/MRI scans.
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Percentage of participants able to complete the PET/MRI examination | Up to 1 year
  Identify the percentage of head and neck cancer patients who are able to successfully complete or partially complete the PET/MRI examination. Responses to a 7 point Likert scale will be analyzed with a chi-squared test.

SECONDARY OUTCOMES:
Changes in staging between PET/CT and PET/MRI | Up to 1 year
  Compare changes in tumor and regional staging between PET/CT and PET/MRI. Responses to a 7 point Likert scale will be analyzed with a chi-squared test.
Feasibility of PET/MRI in radiation treatment planning workflow | Up to 1 year
  Assess the feasibility of PET/MRI in the radiation treatment planning workflow with respect to the adequacy of image quality and image fusion of PET/MRI data with the treatment planning CT, as compared to PET/CT.
Compare conventional MRI pulse sequences to investigational MRI pulse sequences for tumor conspicuity and image quality | Up to 1 year
  Pulse sequences will be assess with Wilcoxon signed rank test.
Compare changes in simulated radiation treatment volume when derived from PET/MRI vs PET/CT (GTV, CTV, PTV) | Up to 1 year
  Differences in simulated radiation treatment planning volumes will be assess with Wilcoxon signed rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Paul M Harari, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- See also: UW Carbone Cancer Center home page — http://www.uwhealth.org/uw-carbone-cancer-center/47424